CLINICAL TRIAL: NCT00173264
Title: Immunologic and Genetic Characteristics of Monoclonal Immunoglobulins in Patient With Tuberculosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700601
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-05

CONDITIONS: Monoclonal Gammopathy; Tuberculosis
MeSH Terms: conditions — Paraproteinemias; Tuberculosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to determine whether the monoclonal protein in patients with tuberculosis and monoclonal gammopathy has anti-tuberculous activity, and whether genes coding their monoclonal proteins show characteristic mutations.

DETAILED DESCRIPTION:
Monoclonal immunoglobulins arise from abnormal proliferation of a single clone of plasma cells. They are composed of a single light and/or heavy chain class, in contrast to polyclonal immunoglobulins. They may occur in malignant lymphoproliferative diseases, such as multiple myeloma, Waldenstrom's macroglobulinemia, lymphoma, chronic lymphocytic leukemia, amyloidosis, or more benign conditions such as monoclonal gammopathy of undetermined significance (MGUS). Recently we have observed monoclonal gammopathy occurring in patients with tuberculosis. Whether tuberculous infection plays a role in the production of monoclonal protein, and whether the monoclonal immunoglobulins possess anti-tuberculous activity are unknown. In the current project we plan to study: (1) whether the monoclonal immunoglobulin developed in patients with tuberculosis reacts with tuberculous antigen (using ELISA), and (2) whether the VH gene sequence analysis of such patient shows different mutation patterns (indicating the presence of intraclonal mutation variation) or not. If there is no intraclonal mutation variation, it suggests that the plasma cell clone is not under current exposure to the mutator, and the production of monoclonal gammopathy is probably not related to tuberculous infection. If, however, the VH gene sequence analysis shows the presence of intraclonal mutation variation, it indicates that the plasma cell clone is continuously under the influence of the mutator. In such case the production of monoclonal protein may be related to tuberculous infection.

ELIGIBILITY:
Inclusion Criteria:

* Monoclonal Gammopathy with Tuberculosis

Exclusion Criteria:

* No

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2005-06; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: LINA LEE, MD,PhD, Principal Investigator — Department of labrotoary medicine,National Taiwan University Hospital
Locations (1):
- Department of Laboratory Medicine, National Taiwan Univeristy Hospital, Taipei, Taiwan